CLINICAL TRIAL: NCT00729157
Title: A Phase II Study of Single Agent Intravenous (IV) VEGF Trap in Patients With Poor Prognostic Recurrent and/or Metastatic Thyroid Cancer After RAI Therapy
Brief Title: Aflibercept in Treating Patients With Recurrent and/or Metastatic Thyroid Cancer That Did Not Respond to Radioactive Iodine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00178; NCI-2009-00178 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MSKCC-08066; CDR0000608163; 08-066 (Other: Memorial Sloan-Kettering Cancer Center); 7508 (Other: CTEP); N01CM62206 (NIH); P30CA008748 (NIH)
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Recurrent Thyroid Gland Carcinoma; Stage III Thyroid Gland Follicular Carcinoma; Stage III Thyroid Gland Papillary Carcinoma; Stage IV Thyroid Gland Follicular Carcinoma; Stage IV Thyroid Gland Papillary Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ziv-aflibercept and fludeoxyglucose F 18) (Experimental): Patients receive aflibercept IV over 1 hour on day 1. Treatment repeats every 14 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients experiencing clear clinical benefit with aflibercept may continue treatment beyond 12 months, at the discretion of the study sponsor. Patients undergo FDG-PET scans at baseline and after 8 weeks of study therapy to evaluate changes in FDG avidity on FDG-PET scan. Blood samples are obtained at baseline and periodically during study for laboratory correlative studies. Samples are examined for pretreatment serum VEGF concentration, thyroglobulin levels (when elevated), serum pharmacokinetics of aflibercept by ELISA, and anti-aflibercept antibodies.
  Interventions: Radiation: Fludeoxyglucose F-18; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Positron Emission Tomography; Biological: Ziv-Aflibercept

INTERVENTIONS:
Radiation: Fludeoxyglucose F-18 — Correlative studies
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Procedure: Positron Emission Tomography — Correlative studies
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Biological: Ziv-Aflibercept — Given IV
  Other Names: AFLIBERCEPT; AVE0005; Vascular Endothelial Growth Factor Trap; VEGF Trap; VEGF Trap R1R2; VEGF-Trap; Zaltrap

SUMMARY:
This phase II trial is studying how well aflibercept works in treating patients with recurrent and/or metastatic thyroid cancer that has not responded to radioactive iodine therapy. Aflibercept may stop the growth of tumor cells by blocking blood flow to the tumor and by carrying tumor-killing substances directly to thyroid cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the radiographic response rate (by RECIST criteria) of IV VEGF Trap after four cycles (approximately 8 weeks) of therapy, as well as the 6-month progression-free-survival (PFS) rate (as part of a composite primary outcome measure), in patients with recurrent and/or metastatic differentiated thyroid carcinoma of follicular cell origin (D-TC-FCO; comprising papillary, follicular, Hurthle cell, and respective variants) not amenable to RAI or curative surgery.

SECONDARY OBJECTIVES:

I. To determine the safety and toxicity profile of IV VEGF Trap in patients with recurrent and/or metastatic TC-FCO. Please see the adverse event table for the specifics for this protocol.

II. To determine the biologic effect of IV VEGF Trap on FDG avidity after four cycles (approximately 8 weeks) of therapy through pre- and post-treatment FDG-PET scans in patients with recurrent and/or metastatic D-TC-FCO.

III. To determine if changes in thyroglobulin concentration after four cycles (approximately 8 weeks) of IV VEGF-Trap therapy correlate with radiographic response after four cycles (approximately 8 weeks) and progression-free-survival at 6 months after start of therapy in patients with recurrent and/or metastatic D-TC-FCO.

IV. To determine if pre-treatment serum VEGF concentration correlates with clinical outcomes after IV VEGF Trap therapy in patients with recurrent and/or metastatic D-TC-FCO.

TERTIARY OBJECTIVES:

I. To determine population pharmacokinetics of IV VEGF Trap for patients with thyroid cancer.

II. To determine whether antibodies to VEGF Trap develop in patients with thyroid cancer.

OUTLINE:

Patients receive aflibercept intravenously (IV) over 1 hour on day 1.

Treatment repeats every 14 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients experiencing clear clinical benefit with aflibercept may continue treatment beyond 12 months, at the discretion of the study sponsor. Patients undergo fludeoxyglucose F 18 (FDG)-PET scans at baseline and after 8 weeks of study therapy to evaluate changes in FDG avidity on FDG-PET scan. Blood samples are obtained at baseline and periodically during study for laboratory correlative studies. Samples are examined for pretreatment serum VEGF concentration, thyroglobulin levels (when elevated), serum pharmacokinetics of aflibercept by ELISA, and anti-aflibercept antibodies.

After completion of study therapy, patients are followed up for 2-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed differentiated thyroid carcinoma of follicular cell origin, including any of the following histologies and their respective variants:

  * Papillary
  * Follicular
  * Hürthle cell
* Must have surgically inoperable and/or recurrent or metastatic disease
* At least one fludeoxyglucose F 18 (FDG)-PET-avid lesion, defined as any focus of increased FDG uptake > normal mediastinal activity with standard uptake variable (SUV) maximum levels ≥ 3, as documented by baseline PET scan
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Progressive disease, defined by ≥ 1 of the following occurring during or after prior treatment (e.g., radioactive isotope [RAI] treatment):

  * Presence of new or progressive lesions on CT scan or MRI
  * New lesions on bone scan or PET scan
  * Rising thyroglobulin level documented by a minimum of 3 consecutive rises, with an interval of > 1 week between each determination
* No known history of brain metastasis
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* ANC ≥ 1,500/mcL
* Platelet count ≥ 75,000/mcL
* WBC ≥ 3,000/mcL
* Total bilirubin ≤ 1.5 times upper limit of normal(ULN)
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN for liver metastases)
* Creatinine ≤ 1.5 times ULNOR creatinine clearance ≥ 60 mL/min
* INR ≤ 1.2 (≤ 1.5 times ULN if on prophylactic-dose anticoagulation)
* Urine protein: creatinine ratio < 1 OR 24-hour urine protein < 500 mg
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 6 months after completion of study therapy
* Documentation of systolic blood pressure ≤150 mm Hg and diastolic blood pressure ≤100 mm Hg
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to other agents used in the study
* No serious or non-healing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess in the past 28 days
* No significant traumatic injury within the past 28 days
* No clinically significant cardiovascular disease, defined as any of the following:

  * Cerebrovascular accident within the past 6 months
  * Myocardial infarction within the past 6 months
  * Coronary artery bypass grafting or unstable angina within the past 6 months
  * NYHA grade III-IV congestive heart failure
  * Canadian Cardiovascular Class grade III or greater angina within the past 6 months
  * Clinically significant peripheral vascular disease within the past 6 months
  * Pulmonary embolism, deep-vein thrombosis, or other thromboembolic event within the past 6 months
  * Uncontrolled coronary artery disease, angina, congestive heart failure, or ventricular arrhythmia requiring acute medical management
  * Myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months
* No evidence of bleeding diathesis or coagulopathy within the past 12 months
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness or social situation that would limit study compliance
* No known HIV positivity
* See Disease Characteristics
* Recovered from prior therapy
* No prior VEGF-targeted antibody therapy (e.g., bevacizumab or aflibercept)
* More than 4 weeks since prior systemic therapy or radiotherapy
* More than 7 days since prior core biopsy
* Up to 1 prior targeted biologic agent (e.g., small-molecule tyrosine kinase inhibitor or histone deacetylase inhibitor) allowed provided treatment was stopped ≥ 4 weeks prior to initiation of therapy on this study
* Up to 1 prior cytotoxic chemotherapy (e.g., doxorubicin hydrochloride) allowed provided treatment was stopped ≥ 4 weeks prior to initiation of therapy on this study
* Prior systemic chemotherapy administered as part of initial definitive treatment (e.g., as a radiation sensitizer or as initial adjuvant therapy) allowed provided treatment was stopped ≥ 3 months prior to initiation of therapy on this study and does not count in the determination of prior targeted or cytotoxic therapy
* At least 2 weeks since prior cyclooxygenase-2 (COX-2) inhibitors, cis-retinoic acid, or complementary medications if given with anti-cancer intent

  * Medications given for a specific clinical indication (e.g., daily aspirin status post myocardial infarction or COX-2 inhibitors at standard anti-inflammatory/pain doses) may be continued based on the clinical judgment of the involved investigator
* Prior RAI therapy allowed provided it was stopped > 3 months prior to initiation of therapy on this protocol and evidence of progression (as defined above) has been documented in the interim

  * A diagnostic study using < 10 mCi of RAI is not considered RAI therapy
* Prior external-beam radiotherapy to index lesions allowed provided there has been documented progression by RECIST criteria and at least 4 weeks have elapsed

  * At least 4 weeks since prior external-beam radiation therapy to non-index lesions
* At least 4 weeks since prior surgery
* Concurrent therapeutic-dose anticoagulants (e.g., warfarin) with PT INR > 1.5 allowed provided that both of the following criteria are met:

  * In-range INR appropriate to the treatment indication (e.g., between 2 and 3 for atrial fibrillation) AND on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* Patients receiving concurrent antihypertensive agents must have documentation of the date of the last change in dosage
* No other concurrent investigational agents
* No major surgical procedure or open biopsy within the past 28 days
* No anticipation of need for major surgical procedures during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-08; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pfister, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ziv-aflibercept and Fludeoxyglucose F 18): Patients receive aflibercept 4mg/kg IV over 1 hour on day 1. Treatment repeats every 14 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients experiencing clear clinical benefit with aflibercept may continue treatment beyond 12 months, at the discretion of the study sponsor. Patients undergo FDG-PET scans at baseline and after 8 weeks of study therapy to evaluate changes in FDG avidity on FDG-PET scan. Blood samples are obtained at baseline and periodically during study for laboratory correlative studies. Samples are examined for pretreatment serum VEGF concentration, thyroglobulin levels (when elevated), serum pharmacokinetics of aflibercept by ELISA, and anti-aflibercept antibodies.
Period: Overall Study
Arm/Group | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18)
Started | 41
Completed | 40
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18)
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival to Determine the 6-month Progression-free-survival (PFS) Rate
Description: Progression-free survival to determine the 6-month progression-free-survival (PFS) rate
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18)
Number analyzed (Participants) | 18
months | 5.4 [1.6 to 30.8]

2. Primary Outcome: Radiographic Response Rate of Aflibercept in Patients With Recurrent and/or Metastatic Thyroid Cancer That Did Not Respond to Radioactive Iodine Therapy
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions & assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + P RMeasurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques (CT, MRI, x-ray) or as ≥ 10 mm with spiral CT scan. All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters). All other lesions (or sites of disease), including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm using spiral CT scan), are considered non-measurable disease. Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, lymphangitis cutis/pulmonis, inflammatory breast disease, abdominal masses (not followed by CT or MRI), & cystic
Time Frame: After 8 weeks of study therapy
Measure: Number; unit: participants
Arm/Group | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18)
Number analyzed (Participants) | 40
participants
  Progression of Disease | 7
  Stable Disease | 33

3. Secondary Outcome: The Safety and Toxicity Profile of IV VEGF Trap in Patients With Recurrent and/or Metastatic TC-FCO
Description: The number of participants, with recurrent and/or metastatic TC-FCO, who experienced adverse events. Please see the adverse event table for the specifics for this protocol.
Time Frame: From the beginning of treatment through 30 days until participant comes off study
Measure: Number; unit: participants
Arm/Group | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18)
Number analyzed (Participants) | 41
participants | 36

4. Secondary Outcome: To Determine the Biologic Effect of IV VEGF Trap on FDG Avidity After Four Cycles (Approximately 8 Weeks) of Therapy Through Pre- and Post-treatment FDG-PET Scans in Patients With Recurrent and/or Metastatic D-TC-FCO.
Description: To determine the biologic effect of IV VEGF Trap on FDG avidity after four cycles (approximately 8 weeks) of therapy through pre- and post-treatment FDG-PET scans in patients with recurrent and/or metastatic D-TC-FCO.
Time Frame: 8 weeks
Measure: Median (95% Confidence Interval); unit: percent of SUVm change
Arm/Group | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18)
Number analyzed (Participants) | 8
percent of SUVm change | .64 [-6.91 to 12.67]

5. Secondary Outcome: Effect of Thyroglobulin Concentration on Progression-free Survival
Description: The change is serum thyroglobulin was measured by the percent change between the baseline value and the lowest value obtained while on treatment.
Time Frame: 6 months
Measure: Median (Full Range); unit: percent change serum thyroglobulin
Arm/Group | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18)
Number analyzed (Participants) | 36
percent change serum thyroglobulin | 0.4 [0 to 90]

6. Other Pre Specified Outcome: To Determine if Pre-treatment Serum VEGF Concentration Correlates With Clinical Outcomes After IV VEGF Trap Therapy in Patients With Recurrent and/or Metastatic D-TC-FCO.
Description: This part is currently under data analysis, therefore, this outcome measure has not been calculatedThis part is currently under data analysis, therefore, this outcome measure has not been calculated.
Time Frame: Baseline-6 months post treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: To Determine if Changes in Thyroglobulin Concentration After Four Cycles (Approximately 8 Weeks) of IV VEGF-Trap Therapy Correlate With Radiographic Response After Four Cycles (Approximately 8 Weeks)
Description: This part is currently under data analysis, therefore, this outcome measure has not been calculated
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18)
Serious Adverse Events (participants affected / at risk) | 24/41
Other Adverse Events (participants affected / at risk) | 36/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18) (N=41)
Cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Cardiac disorder (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Confusion (Psychiatric disorders) | 2 (2)
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Edema: limb (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Hematoma (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 4 (4)
Lymphocyte count decrease (Investigations) | 5 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1)
Neurological disorder (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-cardiac Chest pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Platelet count decrease (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 5 (5)
Renal failure (Renal and urinary disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Thrombotic microangiopathy (Vascular disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ziv-aflibercept and Fludeoxyglucose F 18) (N=41)
Anemia (Blood and lymphatic system disorders) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (11)
Blood bilirubin increased (Investigations) | 4 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 8 (13)
Headache (Nervous system disorders) | 6 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 14 (70)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (5)
Hypertension (Vascular disorders) | 8 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (37)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
INR increased (Investigations) | 2 (27)
Lymphocyte count decreased (Investigations) | 5 (15)
Nausea (Gastrointestinal disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 9 (20)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
White blood cell decreased (Investigations) | 2 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less